CLINICAL TRIAL: NCT03740789
Title: Evaluation of Antiviral Indications and Therapeutic Effect by Liver Biopsy Combined With Clinical Trial Parameters on Chronic HBV Infection With Different Transaminase Levels
Brief Title: Evaluation of Antiviral Indications on Chronic HBV Infection With Different Transaminase Levels
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Yan'an University Affiliated Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2018LSK-146
Record Dates: First submitted 2018-10-28; First posted 2018-11-14 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2018-08

CONDITIONS: Chronic Hepatitis b; ALT
Keywords: Hepatitis B; ALT
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- HBeAg positive: HBeAg positive：group A(ALT≤ULN),group B(ALT 1-2ULN),group C(ALT≥2ULN) and treated subgroup (A1,B1,C1) and untreated subgroup (A2,B2,C2).
- HBeAg negative: HBeAg negative：group A(ALT≤ULN),group B(ALT 1-2ULN),group C(ALT≥2ULN) and treated subgroup (A1,B1,C1) and untreated subgroup (A2,B2,C2).

SUMMARY:
It remains unknown whether antiviral therapy is beneficial for chronic hepatitis B (CHB) with normal or mild ALT.The investigators aim to evaluate the antiviral indications combining liver biopsy and clinical parameters,and further clarify the response indexes of clinical results such as virological, serological, biochemical and histological responses from a retrospective observational cohort study on antiviral therapy in HBeAg positive and negative patients with different ALT levels,especially when ALT lower 2 times upper limit of normal (ULN).

DETAILED DESCRIPTION:
It is estimated that 400 million people worldwide are chronically infected with hepatitis B virus (HBV).Chronic hepatitis B (CHB) often leads to serious health conditions including decompensated liver cirrhosis and hepatocellular carcinoma (HCC). Therefore, the goal of chronic hepatitis B (CHB) therapy is to achieve sustained suppression of HBV replication and remission of liver disease.Clinical CHB management guidelines suggest recommend threshold for antiviral therapy when ALT was more than 2 times ULN.No antiviral drugs are recommended for patients with normal ALT or mildly elevated ALT unless they exhibit symptoms of advanced fibrosis or liver cirrhosis.But chronic HBV infections with normal or mild ALT levels may develop latently into CHB,even cirrhosis and hepatocellular carcinoma (HCC).The ALT level is easily influenced by many factors.Antiviral therapy may still be needed for some HBV patients with normal or mildly abnormal ALT levels. Therefore, the investigator's purpose is to evaluate of antiviral indications and therapeutic effect by liver biopsy and clinical trial parameters on chronic HBV infection with different ALT levels,especially when ALT lower 2 times upper limit of normal (ULN).

ELIGIBILITY:
Inclusion Criteria:All of below

1. Patients with chronic HBV infection,defined as those in whom presence of serum hepatitis B surface(HBsAg) for more than 6 months;
2. All patients had underwent a liver biopsy;
3. All patients signed the informed consent before liver biopsy;
4. No history use of interferon or Nucleoside analogue treatment.

Exclusion Criteria:Any of below

1. Co-infection with hepatitis A virus(HAV),hepatitis C virus(HCV),hepatitis D virus(HDV) hepatitis E virus(HEV) and/or human immunodeficiency virus(HIV);
2. Decompensated cirrhosis;
3. History of hepatocellular carcinoma(HCC);
4. History of liver transplantation;
5. Patient with a history of antiviral treatment;
6. Patient has medical condition that requires concurrent use of systemic prednisolone or other immunosuppressive agent (including chemotherapeutic agent)
7. Patient has one or more additional known primary or secondary causes of liver disease, other than hepatitis B (e.g., alcoholism, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis,alpha-1 antitrypsin deficiency, Wilson's Disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease, etc.)
8. Patient who interrupted antiviral therapy;
9. Patient with incomplete data;
10. Follow up less than 1 year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients underwent a liver biopsy were followed for at least 12 months(range,12-48 months) and follow-up assessments were performed at months 12, 24, 36 and 48.All the patients were detected Serum HBV DNA,HBV markers,including HBsAg,HBsAb,HBeAg,HBeAb,and HBcAb,routine biochemical tests mainly including ALT,AST,TB and ALB,Liver stiffness measurement(LSM) at baseline and endpoint.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Virological response in patients with different ALT levels | at 1 year
  Serum HBV DNA will be summarized and compared between different groups at baseline and follow-up endpoint

SECONDARY OUTCOMES:
Changes in serum HBsAg, HBeAg ,HBeAb ,HBcAb levels between treated and untreated groups | at baseline and 1 year
Proportion of patients with normal alanine aminotransferase(ALT) between treated and untreated groups | at baseline and 1 year
Liver stiffness measurement(LSM) changes between treated and untreated groups | at baseline and 1 year
  LSM response is defined as LSM decrease at least a 1-kilopascal
Proportion of patients with HBsAg loss or seroconversion | at 1 year
(5) Predictive values of HBV DNA,HBsAg and LSM for the antiviral indications of chronic HBV infection with different ALT levels | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yingli He, M.D.,Ph.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The Affiliated Hospital of Yan'an University, Yan’an, Shaanxi, China

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT03740789/Prot_SAP_ICF_000.pdf